CLINICAL TRIAL: NCT06138080
Title: Diagnosing Vesicoureteric Reflux in Children by Direct Isotope Cystography and Contrast Enhanced Voiding Ultrasonography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hanna-Reeta Viljamaa, Principal investigator, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1111
Record Dates: First submitted 2021-10-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: VUR - Vesicoureteric Reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Masking Description: The radiologist and the isotope specialist are not aware of the results of previous VUR investigations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VUR diagnostics (Other)
  Interventions: Diagnostic Test: Contrast-enhanced voiding ultrasonography (CEVUS), Direct isotope cystography

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced voiding ultrasonography (CEVUS), Direct isotope cystography — We have no specific intervention. We investigate different diagnostic modalities of VUR.

SUMMARY:
The purpose of this study is to examine the applicability of contrast enhanced voiding ultrasonography in diagnosing vesicoureteral reflux (VUR) in pediatric patients compared to direct isotope cystography. The aim of the study is to find a modality allowing the accurate diagnosis of VUR and the classification of the degree of VUR with the least possible harm from the examinations.

The investigators recruit 100 under 6 years old patients who have had at least 2 culture positive urinary tract infections. Exluding criteria are abnormal bladder function and posterior uretral valves. The investigators perform direct isotope cystography and contrast enhanced voiding urosonography during the same day to diagnose and grade VUR. The investigators use standardized volume and speed of bladder filling. The examinations are done by a radiologist and an isotope specialist and they are blinded to the result of the other examination.

ELIGIBILITY:
Inclusion Criteria:

* under 6 years old patients who have had at least 2 culture positive urinary tract infections

Exclusion Criteria:

* abnormal bladder function
* posterior uretral valves

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2030-05-15 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accoracy of CEVUS in detecting vesicoureteral reflux | 1 day
  The primary outcome measure of this study is the diagnostic accoracy of CEVUS in detecting vesicoureteral reflux compared to direct isotope cystography, expressed as the sensitivity and specificity of each method

SECONDARY OUTCOMES:
Incidence and severity of adverse effects associated with CEVUS | 1 year
  The secondary outcome measure of this study is the incidence and severity of adverse effects associated with CEVUS as compared to direct isotope cystography.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University hospital, Turku, Finland